CLINICAL TRIAL: NCT01361464
Title: Phase 2 Trial of R115777 in Previously Untreated Older Adults With AML and Baseline Presence of a Specific 2-Gene Expression Signature Ratio
Brief Title: Tipifarnib in Treating Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02589; NCI-2011-02589 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16572; CDR0000699713; 8977 (Other: Moffitt Cancer Center); 8977 (Other: CTEP); P30CA076292 (NIH); N01CM00071 (NIH); U01CA070095 (NIH); N01CM00100 (NIH); NCT01364038 (obsolete NCT alias)
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-02

CONDITIONS: Adult Acute Megakaryoblastic Leukemia; Adult Acute Monoblastic Leukemia; Adult Acute Monocytic Leukemia; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With Maturation; Adult Acute Myeloid Leukemia With Minimal Differentiation; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p22;q23); MLLT3-MLL; Adult Acute Myeloid Leukemia Without Maturation; Adult Acute Myelomonocytic Leukemia; Adult Erythroleukemia; Adult Pure Erythroid Leukemia; Alkylating Agent-Related Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute | interventions — tipifarnib

ARMS (1):
- Treatment (tipifarnib) (Experimental): Patients receive tipifarnib orally twice daily on days 1-21. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Tipifarnib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Tipifarnib — Given PO
  Other Names: R115777; Zarnestra
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well tipifarnib works in treating older patients with acute myeloid leukemia. Tipifarnib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete remission (CR) rate in acute myeloid leukemia (AML) patients prospectively selected for tipifarnib (ZARNESTRA) treatment on the basis of a 2-gene signature (RASGRP1:APTX ratio) in bone marrow aspirates.

SECONDARY OBJECTIVES:

I. To determine the median overall and 1-year survival of patients treated with this regimen II. To determine the median relapse-free survival of patients treated with this regimen.

III. To determine the safety of this regimen in these patients IV. To determine the immunophenotypic expression of RASGRP1 on baseline bone marrow blasts and assess correlation with PCR-based detection.

OUTLINE: This is a multicenter study.

Patients receive tipifarnib orally twice daily on days 1-21. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Bone marrow aspirate and/or biopsy are collected at baseline and on day 28 of course 1 and 2 for RasGRP1 protein expression analysis by qRT-PCR.

After completion of study therapy, patients are followed up every 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated acute myeloid leukemia (AML) (de novo or secondary)

  * No diagnosis of acute promyelocytic leukemia (APL)
* Deemed unsuitable for or refuses standard induction chemotherapy
* RASGRP1:APTX ratio >= 5, through bone marrow screening
* No patients with known leukemic involvement of the central nervous system
* ECOG performance status =< 2
* No WBC >= 30,000/uL (hydroxyurea permitted up to 24 hours prior to initiation of therapy)
* Serum creatinine less than 1.5 times the upper limit of the normal range (ULN) (National Cancer Institute [NCI] Common Toxicity Criteria [CTC] Grade 1)
* Total bilirubin less than 1.5 times ULN (unless the increase is unequivocally due to hemolysis or Gilbert syndrome)
* ALT and AST less than 2.5 times ULN (NCI CTC Grade 1)
* Men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* No symptomatic neuropathy of grade 2 or worse
* No uncompensated disseminated intravascular coagulation (DIC) or uncontrolled bleeding
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to tipifarnib (R115777), such as the imidazole drugs, including clotrimazole, ketoconazole, miconazole, econazole, fenticonazole, isoconazole, sulconazole, ticonazole, or terconazole
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with R115777; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; known HIV-positive patients NOT on antiretroviral therapy AND with a CD4 cell count >= 400/mm^3 are eligible
* No other concurrent cytotoxic or biologic antileukemic therapy
* No patients who are receiving any other investigational agents
* Use of enzyme-inducing anticonvulsants (e.g., phenytoin, fosphenytoin, phenobarbital, primidone, carbamazepine, oxcarbazepine) while taking tipifarnib (R115777) is contraindicated

  * If clinically indicated, subjects may use non-enzyme-inducing anticonvulsants during treatment with R115777

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lancet, Principal Investigator — Moffitt Cancer Center
Locations (7):
- United States (7):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Southeast Phase II Consortium (SEP2C) enrolled participants at 3 cancer centers in the United States. The study opened to accrual on 5/24/2011 and closed to accrual 07/25/2012. Further development of Tipifarnib in acute myeloid leukemia (AML) was terminated after the study failed to meet the primary endpoint.
Groups:
- R115777 Therapy: Each participant will begin R115777 treatment with an orally dosed regimen of 300 mg twice a day (BID) for the first 21 consecutive days of a 28-day cycle.
Period: Overall Study
Arm/Group | R115777 Therapy
Started | 21
Completed | 18
Not Completed | 3
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | R115777 Therapy
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 21
Age, Continuous [Median (Full Range); unit: years] | 75 [66 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate
Description: Complete Remission (CR) rate in Acute Myelogenous Leukemia (AML) patients prospectively selected for R115777R115777 (ZARNESTRA) treatment on the basis of a 2-gene signature (RASGRP1:APTX ratio) in bone marrow aspirates. AML Complete Remission: Bone marrow aspiration - Less than 5% leukemic blasts, Auer rods not detected; Peripheral blood counts - Absolute neutrophil count >/= 1,000/mm^3, Platelet count >/= 100,000/mm^3, Leukemic blasts not present; Blood-product transfusion independence; Absence of extramedullary leukemia.
Time Frame: From first treatment through follow up period, an expected average of 12 months
Population: All evaluable participants
Measure: Number; unit: percentage of participants
Arm/Group | R115777 Therapy
Number analyzed (Participants) | 18
percentage of participants | 11

2. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival is calculated from the first day of R115777 treatment and lasts until the date of death recorded on the case report form (CRF).
Time Frame: From first treatment through follow up period, an expected average of 12 months
Population: All evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | R115777 Therapy
Number analyzed (Participants) | 18
months | 6.6 [4.2 to NA] — Not Reached. Data is through through 12/2012. Updates will be submitted as appropriate.

3. Secondary Outcome: Median 1-Year Survival Rate
Description: Prior to the early discontinuation of the study (for not meeting the primary endpoint of at least 3 CR/CRi after 2 cycles), investigators had planned to calculate one year survival from Kaplan Meier estimates.
Time Frame: 1 year
Population: Evaluable participants at planned study completion date
Arm/Group | R115777 Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Relapse Free Survival
Description: Relapse-free survival is calculated from the date of documentation of complete remission/morphologic complete remission with incomplete blood count recovery (CR/CRi) until disease relapse or death from any cause.
Time Frame: 7 months
Population: All evaluable participants
Measure: Number; unit: participants
Arm/Group | R115777 Therapy
Number analyzed (Participants) | 18
participants | 2

ADVERSE EVENTS:
Time Frame: 19 months
Arm/Group | R115777 Therapy
Serious Adverse Events (participants affected / at risk) | 7/21
Other Adverse Events (participants affected / at risk) | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R115777 Therapy (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (3)
Upper respiratory infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R115777 Therapy (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (11)
Anemia (Blood and lymphatic system disorders) | 4 (5)
Fatigue (General disorders) | 8 (10)
General disorders and administration site conditions - Other (General disorders) | 3 (3)
Chills (General disorders) | 2 (3)
Edema - face (General disorders) | 2 (3)
Fever (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (3)
Pain (General disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 7 (10)
Diarrhea (Gastrointestinal disorders) | 6 (9)
Vomiting (Gastrointestinal disorders) | 6 (8)
Constipation (Gastrointestinal disorders) | 3 (3)
Mucositis - oral (Gastrointestinal disorders) | 2 (2)
Lung infection (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 3 (3)
White blood cell decreased (Investigations) | 7 (9)
Platelet count decreased (Investigations) | 5 (10)
Neutrophil count decreased (Investigations) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6)
Anorexia (Metabolism and nutrition disorders) | 7 (8)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Dizziness (Nervous system disorders) | 4 (6)
Headache (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Confusion (Psychiatric disorders) | 3 (4)
Insomnia (Psychiatric disorders) | 3 (5)
Delirium (Psychiatric disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 3 (4)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 2 (3)

LIMITATIONS AND CAVEATS:
Due to trial not meeting primary endpoint of at least 3 CR/CRi after 2 cycles, accrual was suspended. 1 year survival was not calculated, not relevant in the setting of a median survival of 6.6 months and with study not meeting its primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less